CLINICAL TRIAL: NCT01171456
Title: Early Medical Intervention in Women at Risk for Gestational Diabetes
Brief Title: Early Intervention for Gestational Diabetes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient funding for enrollment of patients. The invesitgators realized the study could not be performed.
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Principal Investigator, Ware Branch, Corporate Med. Director, Women and Newborns, Intermountain Health Care, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1017118
Record Dates: First submitted 2010-07-13; First posted 2010-07-28 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Gestational Diabetes Mellitus
Keywords: GDM; Gestational Diabetes; Diabetes; Pregnancy
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Metformin (Active Comparator)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Administration of Metformin or placebo prior to conception to prevent the onset of GDM.
  Arms: Metformin
Drug: Placebo — Administration of Metformin or placebo prior to conception to prevent the onset of GDM.
  Arms: Metformin Placebo

SUMMARY:
Gestational diabetes (GDM) represents a significant and growing source nationwide of morbidity and mortality for both mothers and infants. Between 5 and 10% of pregnancies are complicated by GDM. Infants exposed in utero to hyperglycemia from GDM have an increased risk of neonatal complications as well as an increased prevalence of a number of chronic diseases, including type 2 diabetes and schizophrenia. Recent research shows that treatment with metformin begun as soon as hyperglycemia is detected in pregnancy is safe and effective. Additional studies demonstrated that metformin is able to decrease the incidence of type 2 diabetes among individuals at risk for this disease. Based upon these findings, the investigators propose to test the hypothesis that metformin therapy for women at risk for gestational diabetes, started prior to conception and before the onset of hyperglycemia, both decreases the incidence of and improves the maternal and neonatal outcomes from GDM.

The investigators intend to conduct a prospective, randomized, double-blind placebo controlled range-finding study to measure the effects of early metabolic intervention with metformin in women at risk for GDM before the commencement of pregnancy or prior to completion of the first trimester. The target sample size for this pilot study is 100 women. The effect size observed will provide preliminary data for a subsequent study which will be sufficiently powered to detect small or moderate effects from early metabolic intervention in women at risk for GDM.

The specific aims of the proposed research consist of the following:

1. Determine whether treating women at risk for GDM with metformin prior to conception and/or completion of the 1st trimester decreases the incidence of GDM at 26 weeks' gestation.
2. Evaluate the effects on maternal and fetal pregnancy outcomes of pre-conception metabolic intervention with metformin in women at risk for GDM.
3. Use these pilot study results to:

   1. identify specific demographic characteristics associated with an intervention effect
   2. calculate effect size for specific outcomes
   3. provide range-finding data for a subsequent study design

Metformin therapy for women at risk for gestational diabetes, started prior to conception and before the onset of hyperglycemia, both decreases the incidence of and improves the maternal and neonatal outcomes from GDM.

ELIGIBILITY:
Inclusion Criteria:

Women delivered >37 weeks gestation in the Intermountain Healthcare Urban Central Region within the last 18 months to ascertain those at risk for GDM in their next pregnancy because of:

* A history of gestational diabetes in their immediately prior pregnancy
* A family history (i.e. type 2 diabetes in a first or second degree relative) of type 2 diabetes
* Delivery of an infant > 4000 gms.
* B.M.I. > 30 six months postpartum
* Hemoglobin A1C > 6.1% six months postpartum

Exclusion Criteria:

Pre-conception exclusion criteria will include any of the following:

* History of >1 miscarriage or fetal demise
* No contraindication to metformin (prior metformin intolerance, metabolic acidosis, GI disease)
* Hypertension (BP >135/85)
* No other endocrine, metabolic, renal, or autommune medical disorders
* Prior preterm birth
* Prior delivery complicated by shoulder dystocia
* Prior delivery complicated by neonatal palsy
* Multifetal pregnancy, including first-trimester embryonic demise of one or more
* Uterine malformations
* Illicit drug or alcohol abuse during current pregnancy
* Intent to deliver elsewhere
* Non-availability for prospective specimen/data collection

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-04; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Effect of metformin versus placebo on the development of GDM | Pre-conception to delivery (at 8 week intervals)

SECONDARY OUTCOMES:
Effects on maternal and fetal pregnancy outcomes of pre-conception metabolic intervention with metformin. | Pre-conception until discharge from hospital after delivery (at 4 week intervals)

CONTACTS AND LOCATIONS:
Overall Officials: Ware Branch, M.D., Principal Investigator — Intermountain Health Care, Inc.
Locations (1):
- Intermountain Medical Center, Murray, Utah, United States